CLINICAL TRIAL: NCT00086021
Title: Acupuncture for the Treatment of Chronic Daily Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23AT001194 (NIH)
Record Dates: First submitted 2004-06-21; First posted 2004-06-22 (Estimated); Last update posted 2007-06-11 (Estimated); Status verified 2007-06

CONDITIONS: Headache Disorders
Keywords: Headache; Acupuncture
MeSH Terms: conditions — Headache Disorders; Headache | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to determine whether acupuncture can reduce pain in long-term headache sufferers.

DETAILED DESCRIPTION:
Acupuncture has been shown to reduce the frequency and severity of some types of headaches, but the efficacy of acupuncture for chronic daily headaches has not been studied. The long-term goals of this study are to reduce the symptoms that are associated with recurrent headaches and to collect data that can be used for future acupuncture studies.

Participants in this study will be randomly assigned to receive 8 weeks of either standard care or ten acupuncture treatments in addition to medical care. Self-report questionnaires will be used to assess headaches and daily pain severity.

ELIGIBILITY:
Inclusion Criteria:

* Ability to communicate in English
* Presence of headache 15 or more days in the past month

Exclusion Criteria:

* Known intracranial mass
* Recent surgery to the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74
Dates: Start 2002-02; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Harvard Medical School, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina